CLINICAL TRIAL: NCT04898894
Title: A Phase I and Expansion Cohort Study of Selinexor and Venetoclax in Combination With Chemotherapy in Pediatric and Young Adult Patients With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Study of Selinexor and Venetoclax in Combination With Chemotherapy in Pediatric and Young Adult Patients With Refractory or Relapsed Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry); AbbVie (Industry); Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SELCLAX; NCI-2021-03435 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2021-05-14; First posted 2021-05-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Leukemia of Ambiguous Lineage in Relapse; Acute Myeloid Leukemia, in Relapse; Refractory Acute Leukemia of Ambiguous Lineage; Refractory Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia, in Relapse; Refractory Acute Myeloid Leukemia; Acute Leukemia of Ambiguous Lineage in Relapse; Refractory Acute Leukemia of Ambiguous Lineage; Pediatric; Young Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute | interventions — venetoclax; selinexor; Cytarabine; fludarabine; fludarabine phosphate; Filgrastim; Granulocyte Colony-Stimulating Factor; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Dose Escalation Phase:
  Venetoclax plus selinexor will initially be given at dose level 1 in combination with intravenous (IV) cytarabine and fludarabine. Dosing of venetoclax and selinexor will be based on tolerability.
  Intrathecal (IT) chemotherapy (IT cytarabine, IT methotrexate, and IT methotrexate/hydrocortisone/cytarabine (MHA) are all acceptable) will be given.
  G-CSF SC may be given.
  Part 1 has been completed and RP2D has been determined to be Dose Level 2. All participants will be treated at Dose Level 2.
  Dose Expansion Phase:
  Two expansion cohorts will be treated at the recommended phase 2 dose (RP2D). Cohort A will include venetoclax-naïve patients, whereas Cohort B will include patients with prior exposure to venetoclax.
  Interventions: Drug: Venetoclax; Drug: Selinexor; Drug: Cytarabine; Drug: Fludarabine; Biological: Filgrastim; Drug: Methotrexate; Drug: methotrexate/hydrocortisone/cytarabine

INTERVENTIONS:
Drug: Venetoclax — Given orally (PO)
  Other Names: Venclextra®; ABT-199
Drug: Selinexor — Given Orally (PO)
  Other Names: KPT-330
Drug: Cytarabine — Given in to the vein (IV) or intrathecal (IT)
  Other Names: Cytosine arabinoside; Ara-C; Cytosar®
Drug: Fludarabine — Given in to the vein (IV) - Because of the ongoing nationwide shortage of fludarabine, this agent may be omitted during the dose expansion phase of the trial.
  Other Names: Fludara®; Fludarabine phosphate; 2-fluoro-ara-AMP
Biological: Filgrastim — Given subcutaneous (SubQ, SC)
  Other Names: G-CSF
Drug: Methotrexate — Given intrathecal (IT)
  Other Names: MTX; amethopterin; Trexall®
Drug: methotrexate/hydrocortisone/cytarabine — Given intrathecal (IT)
  Other Names: ITMHA; Intrathecal triples

SUMMARY:
The purpose of this study is to test the safety and determine the best dose of venetoclax and selinexor when given with chemotherapy drugs in treating pediatric and young adult patients with acute myeloid leukemia (AML) or acute leukemia of ambiguous lineage (ALAL) that has come back (relapsed) or did not respond to treatment (refractory).

Primary Objective

* To determine the safety and tolerability of selinexor and venetoclax in combination with chemotherapy in pediatric patients with relapsed or refractory AML or ALAL.

Secondary Objectives

* Describe the rates of complete remission (CR) and complete remission with incomplete count recovery (CRi) for patients treated with selinexor and venetoclax in combination with chemotherapy at the recommended phase 2 dose (RP2D).
* Describe the overall survival of patients treated at the RP2D.

Exploratory Objectives

* Explore associations between leukemia cell genomics, BCL2 family member protein quantification, BH3 profiling, and response to therapy as assessed by minimal residual disease (MRD) and variant clearance using cell-free deoxyribonucleic acid (DNA) (cfDNA).
* Describe the quality of life of pediatric patients undergoing treatment with selinexor and venetoclax in combination with chemotherapy and explore associations of clinical factors with patient-reported quality of life outcomes.
* Describe the clinical and genetic features associated with exceptional response to the combination of venetoclax and selinexor without the addition of chemotherapy.

DETAILED DESCRIPTION:
This study will include two phases. The dose-escalation phase will characterize the dose-limiting toxicity (DLT) and determine the recommended phase 2 dose (RP2D) of venetoclax plus selinexor with and without chemotherapy. Two expansion cohorts (cohort A, patients without prior exposure to venetoclax; cohort B, patients with prior exposure to venetoclax) will further assess the safety and will explore the efficacy at the RP2D.

Dosing of venetoclax and selinexor will be based on tolerability. Venetoclax will be given orally (po) once daily on days 1 through 21 and selinexor will be given orally (po) starting on days 1, 8, and 15 OR 1, 3, 8, 10, 15, and 17. Beginning on day 16, patients also receive fludarabine phosphate intravenously (IV) daily on days 16-20, cytarabine IV daily on days 16-20, and granulocyte colony-stimulating factor (G-CSF) subcutaneously (SC) daily on days 16-20. G-CSF may be omitted or extended at the discretion of the treating physician. Intrathecal (IT) chemotherapy will be given prior to cycle 1, but may be delayed if clinically indicated. IT cytarabine, IT methotrexate, and IT methotrexate/hydrocortisone/cytarabine (MHA) are all acceptable. Patients without evidence of central nervous system (CNS) leukemia will receive no further IT therapy during cycle 1. Patients with CNS disease will receive weekly IT therapy beginning on day 8, until the cerebrospinal fluid becomes free of leukemia.

Chemotherapy is scheduled to begin on Day 16; however, patients with exceptional responses may, at the discretion of the treating physician, receive chemotherapy (fludarabine and cytarabine) on days 16-20 and continue venetoclax through day 21 and selinexor through day 15 or 17 according to dose level. Alternatively, exceptional responders may continue venetoclax through day 28 and selinexor once or twice weekly according to dose level without chemotherapy and then undergo re-evaluation at day 29. For patients who do not receive chemotherapy on day 16-20, chemotherapy may be omitted completely or may be given on days 30-34 at the discretion of the treating physician.

Patients may receive up to 4 cycles of therapy in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of AML or ALAL and meet the criteria below:

  * Refractory leukemia, defined as persistent leukemia after at least two courses of induction chemotherapy, OR
  * Early relapsed leukemia, defined as the re-appearance of leukemia after the achievement of remission and within one year of diagnosis, OR
  * Relapsed leukemia that is refractory to at least one course of salvage therapy (i.e., therapy given after the relapse has occurred), OR
  * Relapsed leukemia following HCT, OR
  * Second or greater relapse
  * Patients with late first relapses, defined as the re-appearance of leukemia after the achievement of remission and greater than one year of diagnosis, may be enrolled in the dose expansion portion of the study after safety data from the dose escalation portion is available.

Patients must have ≥ 5% blasts in the bone marrow as assessed by morphology or flow cytometry. However, if flow cytometry cannot be performed or if an adequate bone marrow sample cannot be obtained (e.g., in a patient with acute megakaryoblastic leukemia with marrow fibrosis), patients may be enrolled if there is unequivocal evidence of leukemia with ≥ 5% blasts in the blood.

In addition, patients in all categories must not be eligible to undergo curative therapy, such as immediate HCT, because of disease burden, time to identify a stem cell donor, or other reasons.

* Adequate organ function defined as the following:

  * Direct bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * Normal creatinine for age or a calculated creatinine clearance ≥ 30 mL/min/1.73m^2
  * Left ventricular ejection fraction ≥ 40% or shortening fraction ≥ 25%
* Patients must be ≥ 2 years of age and ≤ 30 years old. The upper age limit may be defined by each institution but may not exceed 30 years. Patients treated at St. Jude Children's Research Hospital must be ≤ 24 years old.
* Performance status: Lansky ≥ 50 for patients who are ≤ 16 years old and Karnofsky ≥ 50% for patients who are > 16 years old.
* At least 14 days must have elapsed since the completion of myelosuppressive therapy or hypomethylating agents and the first doses of venetoclax and selinexor.
* At least 24 hours must have elapsed since the completion of low-dose or non- myelosuppressive therapy, such as hydroxyurea, low-dose cytarabine (up to 100 mg/m^2/day), FLT3 inhibitor, or leukapheresis, and the first doses of venetoclax and selinexor.
* For patients who have received prior HCT, there can be no evidence of GVHD and greater than 60 days must have elapsed since the HCT.
* At least 14 days must have elapsed since the completion of any calcineurin inhibitors (e.g. tacrolimus, cyclosporine).
* Patients may not receive strong or moderate CYP3A inducers, such as rifampin, within 3 days of the first dose of venetoclax or during the administration of venetoclax. During the dose-escalation portion of the trial, we discourage the use of strong CYP3A inhibitors (e.g., ketoconazole, itraconazole, voriconazole, posaconazole) within 3 days of the first dose of venetoclax or during the administration of venetoclax. However, if an azole is required for the treatment or prevention of fungal infection during any phase of the trial, venetoclax dosing will be reduced to 60 mg/m^2 (100 mg max) in patients who require treatment with voriconazole and reduced to 40 mg/m^2 (70 mg max) in patients who require posaconazole.

Exclusion Criteria:

* Must not be pregnant or breastfeeding. Male or female of reproductive potential must agree to use effective contraception for the duration of study participation.
* Patients with Down syndrome, acute promyelocytic leukemia, juvenile myelomonocytic leukemia, or bone marrow failure syndromes are not eligible.
* Uncontrolled infection. Patients with infections that are controlled on concurrent anti-microbial agents are eligible.
* Impairment of GI function or GI disease that, in the opinion of the treating physician, may significantly alter the absorption of venetoclax or selinexor.
* History of cerebellar toxicity or cerebellar neurological findings on exam.
* Previous toxicity or hypersensitivity directly attributed to venetoclax.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The recommended phase 2 dose (RP2D) of venetoclax plus selinexor plus chemotherapy. | For each patient, the monitoring time period for dose-limiting toxicity will extend for 35 days from receipt of the first dose of protocol-directed selinexor or venetoclax.
  The primary endpoint is the recommended phase 2 dose (RP2D) of venetoclax plus selinexor plus chemotherapy.
Number of patients treated | 35 days from the receipt of the first dose of protocol-directed selinexor or venetoclax
  A count of the number of patients treated at each dose level during the dose escalation phase will be provided
Number of patients who experience a Non-Hematologic dose limiting toxicity (DLT) during the dose escalation phase | Within 35 days of the first dose of chemotherapy
  A count of the number of patients at each dose level who experience a Non-Hematologic DLT defined as any grade 3 or higher event that occurs within 35 days of the first dose and is at least possibly attributable to study drug administration (venetoclax, selinexor, fludarabine and/or cytarabine).
Number of patients who experience a Hematologic DLT during the dose escalation phase | From the start of chemotherapy up to day 43
  A count of the number of patients at each dose level who experience a Hematologic DLT defined as failure to recover counts (ANC > 500/µl and platelet count > 25,000/µl) by day 43 from the start of chemotherapy unless the delay in count recovery is due to another identifiable factor.

SECONDARY OUTCOMES:
The rates of complete remission (CR) for patients treated with selinexor and venetoclax in combination with chemotherapy at the RP2D. | The final response of each patient will be determined no later than day 42 from the start of chemotherapy.
  CR is defined as bone marrow with < 5% blasts confirmed by flow cytometry, ANC ≥ 500/μL and platelets ≥ 50,000/μL without transfusions, and no evidence of extramedullary disease.
The rates of complete remission with incomplete count recovery (CRi) for patients treated with selinexor and venetoclax in combination with chemotherapy at the RP2D. | The final response of each patient will be determined no later than day 42 from the start of chemotherapy.
  CRi is defined as bone marrow with < 5% blasts confirmed by flow cytometry, ANC < 500/μL or platelets < 50,000/μL without transfusions, and no evidence of extramedullary disease
The overall survival of patients treated at the RP2D. | Survival of each patient will be determined one year from enrollment.
  Overall survival is defined as the time elapsed from protocol enrollment to death, with data for living patients censored at last follow-up. We will report KM estimates with 95% CIs.
The rates of exceptional response for those patients treated during the Dose-escalation phase. | Day 15
  Exceptional Response is defined as patients who have at least 2-log (100-fold) reduction in bone marrow MRD at day 15 compared to bone marrow blast percentage at enrollment.
The rates of exceptional response for those patients treated during the Dose Expansion Phase (Cohort A). | Day 15
  Exceptional Response is defined as patients who have at least 2-log (100-fold) reduction in bone marrow MRD at day 15 compared to bone marrow blast percentage at enrollment.
The rates of exceptional response for those patients treated during the Dose Expansion Phase (Cohort B). | Day 15
  Exceptional Response is defined as patients who have at least 2-log (100-fold) reduction in bone marrow MRD at day 15 compared to bone marrow blast percentage at enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Karol, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (8):
- United States (8):
  - Rady Children's Hospital-San Diego, San Diego, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols

DOCUMENTS (1):
  • Informed Consent Form (2024-12-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04898894/ICF_000.pdf